CLINICAL TRIAL: NCT04441554
Title: High-resolution MRI (7 Tesla) of Foraminal Stenosis and Differentiation of the Degenerated Discovertebral Unit - Comparison with 3 Tesla MRI
Brief Title: High-resolution 7 Tesla MRI of C-spine - Comparison with 3 Tesla MRI
Status: Recruiting | Type: Observational
Sponsor: Balgrist University Hospital (Other)
Responsible Party: Principal Investigator, Reto Sutter, MD, chief of radiology, Balgrist University Hospital
Other Study IDs: R448
Record Dates: First submitted 2020-06-19; First posted 2020-06-22 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-08

CONDITIONS: Magnetic Resonance Imaging; Cervical Spine Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: 7 Tesla MRI — 7 Tesla MRI of cervical spine

SUMMARY:
High-resolution MRI (7 Tesla) of the cervical spine is capable to differentiate osseous spurs from discus-material and better depict the compressed nerve in the neuroforamen compared to 3T MRI.

Provide the surgeon with a detailed high-resolution anatomical image before surgery and potential no need for CT (if the bony anatomy is of crucial importance).

ELIGIBILITY:
Inclusion Criteria:

* Informed consent as documented by signature (Appendix Informed Consent Form)
* >18 years old
* Patients with cervical back pain (radiculopathy) and scheduled surgery for foraminal stenosis or central stenosis or cervical periradicular injection therapy (PRT)

Exclusion Criteria:

* previous surgery
* tumor patients
* pregnancy or breast feeding
* any MRI contra-indications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have undergone a MRI of the spine for clinical indications will be enrolled through consecutive ongoing recruitment in daily clinical practice at Balgrist University Hospital Zurich.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-07-31 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
differentiation of compressed nerves in neuroforamen (7T vs 3T) | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Balgrist University Hospital, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No